CLINICAL TRIAL: NCT06212245
Title: An Open-label Single-arm Clinical Study to Assess the Efficacy and Safety of Inebilizumab in Chinese Adult Patients With Neuromyelitis Optica Spectrum Disorders (NMOSD)
Brief Title: A Clinical Research Study of Inebilizumab in Neuromyelitis Optica Spectrum Disorders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hansoh BioMedical R&D Company (Industry)
Collaborators: Horizon Therapeutics Ireland DAC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-20091-401
Record Dates: First submitted 2023-12-15; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Neuromyelitis Optica Spectrum Disorders
MeSH Terms: conditions — Neuromyelitis Optica | interventions — inebilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inebilizumab (Experimental): Participants will receive IV inebilizumab 300 mg
  Interventions: Drug: Inebilizumab

INTERVENTIONS:
Drug: Inebilizumab — Participants will receive IV inebilizumab 300 mg

SUMMARY:
To assess the efficacy and safety of Inebilizumab in Chinese adult patients with neuromyelitis optica spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have comprehensive understanding of the study content, process and possible adverse reactions, and sign the informed consent forms voluntarily
* Men and women 18 years or older
* Patients with NMOSD diagnosed according to the definition in the Guidelines for the Diagnosis and Treatment of Neuromyelitis Optica Spectrum Disorders in China
* Patients with positive serum anti-AQP4-IgG results at screening
* A documented history of one or more NMOSD acute relapses that required rescue therapy within the last year, or 2 or more NMOSD acute relapses that required rescue therapy within 2 years prior to screening
* Patients with EDSS score of ≤ 7.5 points
* Patients who and whose sexual partner agree to take highly effective method of contraception from screening

Exclusion Criteria:

* Patients who have received any of the following treatments at any time prior to randomization:

  1. Monoclonal antibodies against CD52: such as alemtuzumab, etc.
  2. Total lymphoid irradiation
  3. Bone marrow transplant
  4. T-cell vaccination therapy
* Receipt of rituximab or other B-cell depleting agents (e.g., Belimumab, Telitacicept) within 6 months prior to screening, unless the patient has B-cell counts above the LLN according to the central laboratory;
* Receipt of rituximab or other B-cell depleting agents (e.g., Belimumab, Telitacicept) within 6 months prior to screening, unless the patient has B-cell counts above the LLN according to the central laboratory;
* Patients who have received intravenous injection of immunoglobulin (IVIG) within 1 month prior to randomization;
* Patients who have received immunosuppressant therapy (e.g., cyclophosphamide, methotrexate, mitoxantrone, ciclosporin A, etc.) and biologics (satralizumab, natalizumab, tocilizumab, eculizumab, etc.) within 3 months or 5 half-lives of such drugs (whichever is longer) before randomization;
* Any concomitant disease other than NMOSD that required treatment with oral or IV steroids at doses > 20 mg/day for > 21 days within the 6 months prior to screening;
* Concurrent/previous enrollment in another clinical study involving an investigational treatment within 4 weeks or 5 published half-lives of the investigational treatment, whichever is the longer, prior to enrollment;
* Severe drug allergic history or anaphylaxis to two or more food products or medicine (including known sensitivity to acetaminophen/paracetamol, diphenhydramine or equivalent antihistamine, and methylprednisolone or equivalent glucocorticoid); Known history of allergy or reaction to any component of the investigational product formulation or history of anaphylaxis following any biologic therapy;
* Patients with evidence of alcohol, drug, or chemical abuse, or with history of such abuse within 1 year prior to randomization;
* Female patients who are lactating or pregnant, or plan to become pregnant at any time from signing the informed consent through the study plus 6 months following last dose of investigational product;
* Patients with clinically significant serious active or chronic viral infection, or bacterial infection within 60 days prior to randomization, which requires treatment with anti-infective agents or hospitalization, or might pose an additional risk to the patient in the opinion of the investigator;
* Patients with known history or underlying disease of primary immunodeficiency (congenital or acquired), such as human immunodeficiency virus (HIV) infection or splenectomy, which predisposes the patient to infection;
* Confirmed positive serology results of hepatitis B/C at screening
* Patients with history of malignancy, except squamous or basal cell carcinoma of skin that has been successfully treated with documented success of curative therapy > 3 months prior to randomization;
* Any other conditions that, in the opinion of the investigator, are not suitable for participating in the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-02-25 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with NMOSD attack determined by the investigator | Day 1 (Baseline) through Day 197
  The NMOSD attack is defined as the presence of new or worsening symptom(s) related to NMOSD that meet at least one of the 18 protocol-defined attack criteria. These criteria were developed in conjunction with a panel of disease experts and with Food and Drug Administration input, and were intended to be clinically meaningful, objective, quantifiable, and able to be used worldwide.

SECONDARY OUTCOMES:
Percentage of participants with NMOSD attack determined by the investigator | Day 1 (Baseline) through Day 379
  The NMOSD attack is defined as the presence of new or worsening symptom(s) related to NMOSD that meet at least one of the 18 protocol-defined attack criteria. These criteria were developed in conjunction with a panel of disease experts and with Food and Drug Administration input, and were intended to be clinically meaningful, objective, quantifiable, and able to be used worldwide.
Percentage of Participants With Worsening in Expanded Disability Severity Scale (EDSS) Score | Day 1 (Baseline) through Day 379
  TEDSS and its associated functional system (FS) score provide a system for quantifying disability and monitoring changes in the level of disability over time. EDSS is a scale for assessing neurologic impairment in multiple sclerosis (MS). It consists of 7 FS (visual FS, brainstem FS, pyramidal FS, cerebellar FS, sensory FS, bowel and bladder FS, and cerebral FS) which are used to derive EDSS score ranging from 0 (normal neurological exam) to 10 (death from MS). A negative change from baseline indicates improvement. A participant was considered to have a worsening in overall EDSS score of at least 2 if baseline EDSS score was 0, or at least 1 point if baseline EDSS score is 1 to 5, or at least 0.5 point if baseline EDSS score is 5.5 or more.were measured by MRI of the brain, optic nerve, and spinal cord.
Cumulative Number of Active Magnetic Resonance Imaging (MRI) Lesions | Day 1 (Baseline) through Day 379
  The number of new gadolinium-enhancing lesions and new or enlarging T2 lesions were measured by MRI of the brain, optic nerve, and spinal cord.
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)Laboratory measurements as well as their changes or shift as assessed by CTCAE v5.0 | Day 1 (Baseline) through Day 379
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event is any AE that resulted in death, life threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, is a congenital anomaly/birth defect in offspring of a study participant, is an important medical event that may jeopardize the participant or may require medical intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- IRB of Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No